CLINICAL TRIAL: NCT01612442
Title: Integrated Education Intervention to Improve Infant and Young Child Nutrition and Growth in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: International Development Research Centre, Canada (Other Government)
Responsible Party: Principal Investigator, Agartha Cofie, Principal Investigator (student), McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 290-0310
Record Dates: First submitted 2012-05-27; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Improving Young Child Nutrition
Keywords: complementary feeding; mothers; 6-24 months children; community health volunteers; nutrition education; agricultural education
MeSH Terms: interventions — Nutritional Status; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Integrated education (Experimental)
  Interventions: Behavioral: nutrition and agricultural education
- Control (No Intervention)
- Nutrition education (Experimental)
  Interventions: Behavioral: nutrition education

INTERVENTIONS:
Behavioral: nutrition and agricultural education — Mothers of children aged 6-24 months received monthly nutrition education delivered by community health volunteers and agricultural education delivered by agricultural extension agents, in addition to standard monthly child welfare services delivered by Ghana Health Service
  Arms: Integrated education
Behavioral: nutrition education — Mothers of children aged 6-24 months received monthly nutrition education delivered by community health volunteers in addition to standard child growth monitoring services provided by the Ghana Health Service.
  Arms: Nutrition education

SUMMARY:
In Ghana the level of malnutrition is high among children below five years of age, particularly in rural areas. The objective of the study was to investigate the effects of an education intervention aimed at addressing poor complementary feeding (CF) practices on the food intakes and growth of young children in the Upper Manya Krobo district of Ghana.

Interviews and focus group discussions involving community health and agricultural workers, as well as caregivers of children 6-24 months old were conducted to investigate the facilitators and challenges to optimal CF practices and education on CF. The trials of improved practices (TIPs) method was used to test the feasibility and acceptability of potential education messages among mothers of young children (6-24 months) living in the study area. Child welfare clinic centers in the area were randomly assigned to one of three groups which were control, nutrition education and integrated education. Mothers of children 6-24 months in the integrated education group received monthly nutrition education from community health volunteers and agricultural education from agricultural extension agents for six months in addition to standard monthly child growth monitoring services from community health nurses. Mothers in the nutrition education group received monthly nutrition education from community health volunteers for six months in addition to standard care. Mothers of 6-24 months in the control group received only the standard monthly child monitoring services. The effects of the educational intervention on maternal knowledge on optimal complementary feeding, as well as food intakes and growth of young children were determined among 367 mother-child dyads over a period of at least six months. The study hypothesised that mothers receiving the education would have improved knowledge on good complementary feeding practices compared to those in the control group. The study also hypothesised that young children in the integrated education would have better nutrient intakes and growth compared those in the nutrition education and control groups, and those in the nutrition education group would have better nutrient intakes and growth than the children in the control group.

From the interviews and focus group discussions, reported initiation of CF was satisfactory, while other reported practices such as the addition of animal source foods, vegetables and fruits to young children's diet were found to be sub-optimal. Poverty and maternal time constraints were identified as the main challenges of optimal complementary feeding, while farming was seen as a facilitator. Lack of education materials, language barrier, maternal time constraints and lack of in-service training for health workers were the main challenges to education on complementary feeding. From the TIPS study, mothers expressed their willingness to improve the diets of their 6-24 months old children by adding or increasing the amount of animal source foods, dark-green leafy vegetables and fruits, as well as increasing feeding frequency daily. However, availability and affordability of protein-rich foods like animal source foods, groundnut paste and soya beans powder was a challenge for some mothers.

The intervention did not lead to a significant improvement in maternal knowledge on complementary feeding practices. However, it showed a tendency to reverse a general decreasing trend in knowledge among mothers on appropriate complementary feeding practices in the study area. Significantly more children in the integrated education group consumed animal source foods compared those in the other two groups when compared at nine months after baseline. However, the intervention did not improve the general nutrient intakes and growth of the young children in the study area.

ELIGIBILITY:
Inclusion Criteria:

* child aged 6-11 months old and attending monthly growth monitoring clinic
* mother and child living in the study area

Exclusion Criteria:

* birth defects which results in difficulty in feeding of child

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 367 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
growth (change in weight and length) | 9 months

SECONDARY OUTCOMES:
maternal nutrition knowledge | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Marquis, PhD, Study Director — McGill University
Locations (1):
- Upper Manya Krobo district, Assesewa, Eastern Region, Ghana